CLINICAL TRIAL: NCT00636480
Title: Preoperative Skin Preparation Evaluation of One Test Product With a Positive and a Negative Control
Brief Title: Preoperative Skin Preparation Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 070921-103
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Topical Antisepsis
Keywords: Antimicrobial; Antisepsis
MeSH Terms: interventions — chlorhexidine gluconate; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHG 2%-26 ml (Experimental): Chlorhexidine gluconate in an aqueous base, 26 ml applicator
  Interventions: Drug: Chlorhexidine gluconate
- ChloraPrep 26 ml (Active Comparator): ChloraPrep One-Step 26 ml Active drug contains chlorhexidine gluconate and alcohol
  Interventions: Drug: ChloraPrep One Step
- Sterile Saline (Placebo Comparator): Sterile salt water administered topically.
  Interventions: Drug: Sterile saline

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Chlorhexidine gluconate (2% w/v) in an aqueous base, 26 ml applicator. Active drug contains alcohol and the placebo contains no drug. Administered topically.
  Other Names: ChloraPrep AQ
  Arms: CHG 2%-26 ml
Drug: ChloraPrep One Step — Administer topically
  Other Names: Chlorhexidine gluconate 2% w/v and 70% v/v isopropyl alcohol
  Arms: ChloraPrep 26 ml
Drug: Sterile saline — 0.9% NaCl solution
  Other Names: Physiologic saline (0.9% NaCl)
  Arms: Sterile Saline

SUMMARY:
Determine the antimicrobial properties of a proposed new product and an already approved product and a placebo (no drug). Study will be conducted using methods dictated by the FDA.

DETAILED DESCRIPTION:
Determine the antimicrobial properties of a proposed new product and an already approved product and a placebo (no drug). Study will be conducted using methods dictated by the FDA.

This study uses topical sampling from the abdomen and the groin on intact skin and evaluates the germs left on the skin after treatment with the proposed new product, the currently approved product and the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Free of dermatoses, cuts, lesions, or other skin disorders on or around the test sites; no exposure to topical or systemic antimicrobials, antibiotics, or steroids (other than contraceptives, for the fourteen (14) day pre-test conditioning period and must agree to abstain from these materials until completion of the study

Exclusion Criteria:

* Exposure of test sites to antimicrobial agents, medicated soaps, medicated shampoos, or medicated lotions,
* Use of biocide-treated pools or hot tubs, use of tanning beds, or sunbathing during the fourteen(14) day pre-test conditioning period or during the test period;
* Exposure of the test sites to strong detergent, solvents, or other irritants during the fourteen (14) day pre-test conditioning period or during the test period;
* Use of systemic or topical antibiotic medications, steroid medications other than contraceptives, or any other product known to affect the normal microbial flora of the skin during the fourteen ()14) day pre-test conditioning period or during the test period;
* Know of allergies to vinyl, latex (rubber), alcohols, metals, inks, or tape adhesives, or to common antibacterial agents found in soaps, lotions, or ointments, particularly chlorhexidine gluconate, and/or isopropyl alcohol;
* A medical diagnosis of a physical condition, such as a current or recent severe illness, asthma, diabetes, hepatitis, an organ transplant, any immunocompromised conditions such as AIDS (or HIV positive), mitral valve prolapse, or a requirement to take antibiotics prior to dental procedures;
* Pregnancy, plans to become pregnant within the pre-test and test periods of the study, or nursing a child;
* Any active skin rashes or breaks in the skin of the test sites;
* A currently active skin disease or inflammatory skin condition, including contact dermatitis; showering or bathing within the seventy-two (72) hour period prior to sampling; participation in another clinical study in the past thirty (30) days or current participation in another clinical study;
* Any medical condition or use of any medications, that, in the opinion of the Study Director, should preclude participation;
* Unwillingness to fulfill the performance requirements of the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
3.0 log10 reduction in CFU/cm2 on inguinal sites, and 2.0 log10 reduction in CFU/cm2 on abdominal sites | 10 minutes and 6 hours after application of test solutions

CONTACTS AND LOCATIONS:
Overall Officials: Daryl S Paulsen, PhD, Principal Investigator — President and CEO
Locations (1):
- BioScience Laboratories, Bozeman, Montana, United States